CLINICAL TRIAL: NCT02314611
Title: Post Market Clinical Follow-Up Study Protocol for PROFEMUR® Gladiator HA Coated Modular Femoral Stems
Status: Terminated | Type: Observational
Why Stopped: The primary reason for this study was to collect safety and performance data to meet regulatory requirements. However, these requirements have changed over time. Our recentassessment has determined that now there is sufficient data on this product.
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-LJH-002D
Record Dates: First submitted 2014-12-08; First posted 2014-12-11 (Estimated); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Joint Disease
Keywords: osteoarthritis; avascular necrosis; ankylosis; protrusio acetabuli; painful hip dysplasia; rheumatoid arthritis; correction of functional deformity; revision procedures
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Osteonecrosis; Ankylosis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PROFEMUR® Gladiator HA Coated Stem: Single study group previously implanted with a primary PROFEMUR® Gladiator HA Coated Modular Femoral Stem (HA = Hydroxyapatite)
  Interventions: Device: PROFEMUR® Gladiator HA Coated Modular Femoral Stem

INTERVENTIONS:
Device: PROFEMUR® Gladiator HA Coated Modular Femoral Stem — Total Hip Arthroplasty (THA) using PROFEMUR® Gladiator HA Coated Modular Femoral Stem
  Other Names: Primary hip replacement device

SUMMARY:
MicroPort Orthopedics (MPO) is conducting this post market clinical follow-up (PMCF) study to evaluate the safety and efficacy of its total hip arthroplasty (THA) and resurfacing components marketed in the European Union (EU). These types of studies are required by regulatory authorities for all THA and resurfacing devices that do not have medium to long-term clinical evidence available at the time of gaining approval to market in the EU. This study has been designed in accordance with the medial device directives (MEDDEV) 2.12/2 rev 2.

ELIGIBILITY:
Inclusion Criteria:

* Subject has undergone primary THA for any of the following:
* Non-inflammatory degenerative joint disease such as osteoarthritis, avascular necrosis, ankylosis, protrusio acetabuli, or painful hip dysplasia;
* Inflammatory degenerative joint disease such as rheumatoid arthritis; or
* Correction of functional deformity
* Subject is implanted with the specified combination of components
* Subject is willing and able to complete required study visits or assessments

Previously implanted bilateral subjects can have both THAs enrolled in the study provided: 1) the specified combination of components were implanted in both, 2) all other aspects of the Inclusion/Exclusion Criteria are satisfied, 3) enrollment does not exceed the subject count specified in the Investigator Agreement, and 4) the subject agrees to a second Informed Consent document specific to the second THA. Prospective enrollment of a previously unimplanted hip is not permitted in this study.

Exclusion Criteria:

* Subjects skeletally immature (less than 21 years of age) at time of primary THA surgery
* Subjects currently enrolled in another clinical study which could affect the endpoints of this protocol
* Subjects unwilling to sign the Informed Consent document
* Subjects with substance abuse issues
* Subjects who are incarcerated

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been previously implanted with a PROFEMUR® Gladiator HA Coated Modular Femoral Stem
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2023-11 (Actual)

PRIMARY OUTCOMES:
Component Survivorship | 10 years post-operative
  The primary objective of this study is to estimate survivorship of all components at specified intervals out to 10 years follow-up.

SECONDARY OUTCOMES:
Patient functional outcomes (hip specific) | 5 months, 1, 2, 5, 7, and 10 years beginning with first available follow-up interval
  To characterize total functional scores, as assessed by Hip disability and Osteoarthritis Outcome Scores (HOOS)
Patient functional outcomes (quality of life) | 5 months, 1, 2, 5, 7, and 10 years beginning with first available follow-up interval
  To characterize total functional scores, as assessed by EQ-5D-3L scores

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Van Overschelde, MD, Principal Investigator — Algemeen Ziekenhuis Maria-Middelares (Gent, Belgium)
Locations (1):
- Medisch Centrum Latem (outpatient clinic associated with AZ Maria-Middelares), Sint-Martens-Latem, Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No